CLINICAL TRIAL: NCT02947126
Title: Multilevel Models of Therapeutic Response in the Lungs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tim Corcoran (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Tim Corcoran, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PRO15070376; 1U01HL131046-01 (NIH)
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; mucociliary clearance; CFTR
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic; Sodium Chloride; Pentetic Acid; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cystic Fibrosis (HS, IS) (Experimental): CF subjects: ages 12 or older with a diagnosis of cystic fibrosis as determined by sweat test or genotype and clinical symptoms who are clinically stable as determined by a physician co-investigator. Subjects receive HS dose on first imaging day and IS dose on the second imaging day,
  Indium-DTPA (1.5 mCi), Technetium sulfur colloid (8mCi), Inhaled isotonic saline (4ml), Inhaled Hypertonic Saline (4ml)
  Interventions: Drug: Hypertonic Saline; Drug: Isotonic Saline; Drug: Indium-DTPA; Drug: Technetium Sulfur Colloid
- Cystic Fibrosis (IS, HS) (Experimental): CF subjects: ages 12 or older with a diagnosis of cystic fibrosis as determined by sweat test or genotype and clinical symptoms who are clinically stable as determined by a physician co-investigator. Subjects receive IS dose on first imaging day and HS dose on the second imaging day.
  Indium-DTPA (1.5 mCi), Technetium sulfur colloid (8mCi), Inhaled isotonic saline (4ml), Inhaled Hypertonic Saline (4ml)
  Interventions: Drug: Hypertonic Saline; Drug: Isotonic Saline; Drug: Indium-DTPA; Drug: Technetium Sulfur Colloid
- Parents of CF subjects (Experimental): Ages 18 and older, biological parent of a CF patient who is also enrolled in the study
  Indium-DTPA (1.5 mCi), Technetium sulfur colloid (8mCi), Inhaled isotonic saline (4ml)
  Interventions: Drug: Isotonic Saline; Drug: Indium-DTPA; Drug: Technetium Sulfur Colloid
- non CF controls (Experimental): Ages 18 and older with no history of lung disease
  Indium-DTPA (1.5 mCi), Technetium sulfur colloid (8mCi), Inhaled isotonic saline (4ml).
  Interventions: Drug: Isotonic Saline; Drug: Indium-DTPA; Drug: Technetium Sulfur Colloid

INTERVENTIONS:
Drug: Hypertonic Saline — Inhaled 7% Hypertonic saline
  Arms: Cystic Fibrosis (HS, IS); Cystic Fibrosis (IS, HS)
Drug: Isotonic Saline — Inhaled 0.9% Isotonic saline
Drug: Indium-DTPA — Inhaled Indium 111 DTPA
Drug: Technetium Sulfur Colloid — Inhaled Technetium99m sulfur colloid

SUMMARY:
When developing new medications for lung diseases like Cystic Fibrosis (CF), scientists perform lab experiments using cells from the airways, physiology studies of how the lungs change when a drug is given, and clinical studies to determine how drugs affect overall health. The investigators of this study are seeking to develop computer models that will predict how patients will respond to drugs by just doing lab studies on cell samples from their noses. Such models would allow for medications to be developed more rapidly for all patients and allow treatments to be personalized as well. In order to develop these computer models a series of tests will be performed on patients who have CF. Tests will include sampling cells from the nose and measuring lung physiology using a combination of different imaging, breathing, and other studies performed both before and after participants take a therapy. Similar tests will be performed on people who do not have CF, and on the parents of the CF participants who carry a single CF gene because this will provide information on how specific genes might affect CF lung disease.

DETAILED DESCRIPTION:
The goal of this research is to develop a series of interconnected models of therapeutic response in the diseased lung, focused primarily on Cystic Fibrosis (CF), that will ultimately provide a means for predicting in vivo response based on patient-specific in vitro testing, allowing for the optimization and personalization of therapies. Investigators use both human bronchial epithelial (HBE) and more recently human nasal epithelial (HNE) cell cultures to study CF pathophysiology. The investigators performing this study have also developed functional imaging biomarkers in the lung that provide organ level quantification of CF lung physiology (mucociliary clearance and airway liquid absorption), and, more recently, in silico systems models of lung physiology at both the cell and organ level. The in silico models provide a framework of differential equations that describe how basic physiological processes interact and contribute to experimental outcomes. Their use allows these mechanisms to be more specifically differentiated. Here the investigators propose to link in vitro and in vivo response by sampling and culturing HNE cell cultures from both non-CF and CF subjects who will also perform a series of physiological assessments, including functional imaging scans. The in silico models will facilitate linking therapeutic studies in cells to therapeutic outcomes in patients.

1. CF PATIENTS will perform 2 study days.

   Study day 1 will include:
   1. nasal potential difference measurements
   2. pulmonary function testing
   3. inert gas washout testing
   4. urine pregnancy testing
   5. nasal cell sampling
   6. nuclear MCC/ABS scan (to include inhalation of isotonic or hypertonic saline - randomized order)
   7. blood draw for CFTR genotyping if not already available.

   Study day 2 will include
   1. pulmonary function testing
   2. urine pregnancy testing
   3. nuclear MCC/ABS scan (to include inhalation of isotonic or hypertonic saline - randomized order)
2. PARENTS OF ENROLLED CF patients who choose to participate will perform 1 study day which will include:

   1. nasal potential difference measurements
   2. pulmonary function testing
   3. inert gas washout testing
   4. urine pregnancy testing
   5. nasal cell sampling
   6. nuclear MCC/ABS scan (to include inhalation of isotonic saline)
   7. a single blood sample drawn for CFTR genotyping.
3. HEALTHY CONTROLS will perform 1 screening and 1 study day which will include:

   1. pulmonary function testing
   2. inert gas washout testing
   3. urine pregnancy testing
   4. nasal cell sampling
   5. nuclear MCC/ABS scan (to include inhalation of isotonic saline)
   6. a single blood sample drawn for CFTR genotyping (at screening).

ELIGIBILITY:
Cystic Fibrosis Subjects: Inclusion Criteria

* Ages 12 or older
* Diagnosis of cystic fibrosis as determined by sweat test or genotype
* Clinically stable as determined by a physician co-investigator

Cystic Fibrosis Subjects: Exclusion Criteria

* Smokers or users of electronic cigarettes
* FEV1%p <30% of predicted
* Nursing, pregnant or unwilling to test for pregnancy
* Intolerant to hypertonic saline
* Unable or unwilling to discontinue hypertonic saline, Pulmozyme, and long acting bronchodilators for 24 hrs before testing and short acting bronchodilators on testing days.

CF parents: Inclusion Criteria

* Ages 18 and older
* Biological parent of a CF patient who is also enrolled in the study

CF parents: Exclusion Criteria

* Smokers or users of electronic cigarettes
* FEV1%p <30% of predicted
* Nursing, pregnant or unwilling to test for pregnancy
* Unwilling to discontinue long acting bronchodilators for 24 hrs before testing and short acting bronchodilators on testing days.
* Unwilling to perform CFTR genotyping.

Healthy controls: Inclusion Criteria

* Ages 18 and older
* No history of lung disease

Healthy Controls: Exclusion Criteria

* Smokers or users of electronic cigarettes
* FEV1%p <70% of predicted
* Nursing, pregnant or unwilling to test for pregnancy
* Carriers of known disease causing CFTR mutations
* Unwilling to perform CFTR genotyping.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Mucociliary Clearance | 80 minutes
  Clearance rate of Technetium sulfur colloid from the lungs
DTPA absorption rate | 80 minutes
  DTPA absorption rate from the lungs (difference between total In-DTPA clearance rate and mucociliary clearance rate)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Corcoran, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Publication describing outcomes — https://openres.ersjournals.com/content/8/4/00382-2022